CLINICAL TRIAL: NCT03795389
Title: A Multi-Center Open-label Investigation to Assess the Pharmacokinetics, Safety and Tolerability of DM199 in Patients With Diabetes Mellitus and Chronic Kidney Disease
Brief Title: Study to Assess PK, Safety and Tolerability in Patients With DM and CKD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DiaMedica Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DM199-2018-001
Record Dates: First submitted 2019-01-03; First posted 2019-01-07 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2019-07

CONDITIONS: Chronic Kidney Disease; Chronic Kidney Disease, Stage 3 (Moderate); Chronic Kidney Disease, Stage 4 (Severe); Diabetes
Keywords: Diabetes; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Lymphoma, Follicular; Diabetes Mellitus | interventions — DM199

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 3.0 µg/kg SC, single dose (Experimental): n=8, study group of T1D or T2D with stage 3 CKD. separate n=8 of study group with T1D or T2D with CKD stage 4).
  Interventions: Drug: DM199
- 5.0 µg/kg SC, single dose (Experimental): n=8, study group of T1D or T2D with stage 3 CKD.
  Interventions: Drug: DM199
- 8.0 µg/kg SC, single dose (Experimental): n=8, study group of T1D or T2D with stage 3 CKD.
  Interventions: Drug: DM199

INTERVENTIONS:
Drug: DM199 — Single SC dose

SUMMARY:
An open-label, phase IB, multi-center study evaluating DM199 in subjects with Type 1 Diabetes or Type 2 Diabetes and Stage 3 or 4 Chronic Kidney Disease. The primary objectives of this study are to evaluate safety, tolerability, and PK profile of DM199 in these subjects.

DETAILED DESCRIPTION:
The study evaluates the safety, tolerability, and PK profile of DM199 in subjects with T1D or T2D and with Stage 3 or Stage 4 CKD. Additionally, this study evaluates urine concentrations of KLK1 pre and post dose.

Cohort 1: Subjects with T1D or T2D and Stage 3 CKD will be administered one of three DM199 doses: 3.0 ug/kg or 5.0 ug/kg or 8.0 ug/kg single SC dose. Cohort 2: Subjects with T1D or T2D and Stage 4 CKD will be administered a single 3.0 µg/kg single SC dose. Secondary and exploratory study objectives include collection and analysis of vital signs, biomarkers, eGFR, blood glucose, and ECG's.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to provide informed consent for study participation.
* Subject is ≥ 18 years of age.
* Subject has an established diagnosis of T1D or T2D as determined by medical evaluation at screen.
* Subjects A1c <9.8%
* Subject is clinically stable with respect to underlying renal impairment and diabetes, as assessed by the Investigator's medical evaluation.
* Subject has been diagnosed with Stage 3 CKD as defined by eGFR (MDRD) between 30 - <60 or Stage 4 as defined by eGFR <30 (not on dialysis) at screening.
* Subject has a body mass index (BMI) between 18 to 45 kg/m2 (inclusive).

Exclusion Criteria:

* Subject has positive drug test for drugs of abuse and/or positive alcohol breath test at screening and Day 0.
* Subject is unable or unwilling to comply with protocol requirements, including assessments, tests, and follow-up visits.
* Subject has a history of significant allergic diathesis such as urticaria, angioedema, or anaphylaxis.
* Subject has had any live vaccination ≤ 3 months prior to enrollment or will require vaccination during the study.
* Subject must not be taking an ACEi medication for 5 half-lives prior to study drug administration and for 5 days post study drug administration.
* Subject is unwilling or unable to limit smoking to ≤ 10 cigarettes per day (or other products that contain nicotine limited to < 200 mg of nicotine/day) during the study participation period.
* Subject has a current malignancy or active malignancy ≤ 3 years prior to enrollment except basal cell or squamous cell carcinoma of the skin or in situ cervical cancer that has undergone potentially curative therapy and ≥ six months have elapsed since the procedure.
* Subject has an active infection at the time of enrollment, and/or a history of clinically significant acute bacterial, viral, or fungal systemic infections that required systemic treatment in the last four weeks prior to enrollment.
* Subject has known medical history of alpha 1-antitrypsin deficiency (α1-antitrypsin deficiency).
* Subject has serological evidence of human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or anti-hepatitis C virus (Anti-HCV) at screen.
* Subject is pregnant or nursing or is planning a pregnancy during the study period.
* Subject is male or female of childbearing potential, is participating in sexual activity that could lead to pregnancy and is unable or unwilling to practice medically effective contraception during the study.
* Subject has received any investigational drug or device within 14 days (or 5 half lives, whichever is longer) prior to study drug administration on Day 1
* Subject has renal artery stenosis as determine at screen with medical history.
* Subject has hypotension as defined by systolic blood pressure ≤ 90 and diastolic blood pressure ≤ 60 mmHg.
* Subject has Proteinuria: PCR>2000mg/gm (spot testing).
* Subject does not have adequate venous access for blood sampling.
* Subject has any other medical condition which, in the opinion of the Investigator, will make participation medically unsafe or interfere with the study results.
* Subject has any other clinically significant abnormalities in laboratory test results at screening that would, in the opinion of the Investigator, increase the subject's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data.
* Subject has any of the following conditions as determined by ECG or medical record:

  * Any significant arrhythmia or conduction abnormality, which, in the opinion of the Investigators and Medical Monitor, may interfere with the safety of the subject.
* Subject is taking Cimetidine, St. John's Wort, or any other herbal or probiotic supplement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2019-07-21 (Actual); Study Completion 2019-07-21 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by incidence, severity, and causality of adverse events | 11 days
Tolerability as assessed by incidence and severity of AEs | 11 days
plasma measurements of DM199 | 11 days
  as measured in the three different dosing groups; 3.0 ug/kg, 5.0 ug/kg, and 8.0 ug/kg.
DM199 urine concentrations of KLK1 | 11 days
  urine KLK1 will be measured pre and post study drug administration.

SECONDARY OUTCOMES:
C Reactive protein (CRP) | 11 days
Matrix Metalloproteinase-9 (MMP-9) | 11 days
Vascular Endothelial Growth Factor (VEGF) | 11 days
Nitric Oxide (NO) | 11 days
Serum creatinine | 11 days
Cystatin C | 11 days
neutrophil gelatinase-associated prostaglandin E2 | 11 days
Urine Kidney Injury Molecule-1 (Kim1) | 11 days

OTHER OUTCOMES:
serum creatinine | 11 days
Blood glucose | 11 days

CONTACTS AND LOCATIONS:
Overall Officials: Harry Alcorn, Pharm.D., Study Director — DiaMedica Inc.
Locations (3):
- United States (3):
  - Clinical Pharmacology of Miami, Hialeah, Florida
  - Orlando Clinical Research Center Inc, Orlando, Florida
  - Prism Research, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No